CLINICAL TRIAL: NCT01569932
Title: Cognitive and Functional Changes With Chemotherapy in Adult Cancer
Brief Title: Cognitive Changes in Adult Cancer Survivors
Acronym: CFCC
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Jay F. Piccirillo, MD, Professor of Otolaryngology, Director of Clinical Outcomes Research Office, Washington University School of Medicine
Other Study IDs: 201105082
Record Dates: First submitted 2012-03-07; First posted 2012-04-03 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Effects of Chemotherapy; Cognitive Impairment
Keywords: chemobrain, chemotherapy, cognitive impairments, fcMRI, neurocognitive Assessments
MeSH Terms: conditions — Cognitive Dysfunction; Chemotherapy-Related Cognitive Impairment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- chemotherapy: Patients will be assessed both before and after they undergo treatment with chemotherapy.

SUMMARY:
This study will document the cognitive (mental) and functional abilities of newly diagnosed cancer patients. The study will also examine the changes in cognitive and functional abilities during and after chemotherapy (your cancer treatment).

A comprehensive set of questionnaires and tasks, or assessments, have been put together in order for doctors and nurses to learn more about the day to day functioning of newly diagnosed adult cancer patients. The investigators would also like to follow up with the same adult patients, during and following completion of their cancer treatment, to learn about the kinds of treatments they received and how their cognitive status and level of participation in activities of daily living has changed. With follow-up assessments, doctors and nurses can learn more about the complications or health problems that adult patients may experience as a result of undergoing cancer therapy. This is a study involving two visits. The first visit occurs within two weeks before starting your cancer therapy, specifically chemotherapy. The second visit occurs within two weeks of completing your chemotherapy.

DETAILED DESCRIPTION:
Chemotherapy is increasingly used in the management of various cancers. There are reports in the literature of chemotherapy-induced cognitive impairments ranging from deficits in memory and attention to slowed information-processing and deficiencies in executive function, including planning and problem-solving. These deficits have been shown to affect work-place productivity and social role-functioning which present significant public health risks in an era of increased chemotherapy usage. However, previous studies investigating cognitive deficits after chemotherapy have mainly used neurocognitive assessments, which are limited in their utility for clinical diagnosis due to their likelihood for practice effects and low sensitivity for detecting subtle cognitive changes that may be functionally relevant to the patient.

Resting-state functional connectivity magnetic resonance imaging (fcMRI) is a sensitive test that measures resting-state neural network connectivity, reflecting the integrity between functionally-related brain regions. fcMRI has been used to delineate cortical neural networks involved in a variety of cognitive domains, including memory, and attention. The investigators believe that fcMRI will be more sensitive than neurocognitive tests alone for investigating chemotherapy-induced cognitive changes. The goal of this novel study is to use fcMRI to investigate cognitive changes after chemotherapy in an attempt to understand the currently unknown neurobiological mechanisms associated with this phenomenon.

This prospective study will investigate the presence of cognitive deficits after chemotherapy in cancer patients by assessing changes in three fcMRI-defined neural networks involved in cognition. The three networks include (1) Dorsal Frontal Attention network (2) "Default" network and (3) Cognition "Core" control network. Sixteen cancer patients scheduled for chemotherapy will undergo fcMRI of the brain and neurocognitive testing within two weeks before and after chemotherapy. Comparisons between time-points will establish the effect of chemotherapy on cognition.

Results obtained from this study in cancer patients will provide insight into the mechanisms underlying the development of chemotherapy-induced cognitive deficits. Knowledge of the development of chemotherapy-induced cognitive deficits will enhance positive outcomes by allowing practitioners and patients to be better informed of the potential cognitive consequences to anticipate. With patients equipped with such information before starting cancer treatment, they will be better able to manage their affairs and daily activities in such a way that allows them to maintain productive living through their course of cancer and its treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 40 years of age or older
* Subjects must be able to read, write and speak English fluently
* Treatment with a chemotherapy regimen that contains 5-fluorouracil or a platinum-based drug.
* Breast cancer subjects must be newly diagnosed with invasive lobular or ductal cancer (stages II and III)
* Head and Neck cancer subjects must be newly diagnosed with locally-advanced squamous cell carcinoma of the head and neck in oropharyngeal, hypopharyngeal and laryngeal sites (stages III and IV)
* Ovarian, fallopian tube, or primary peritoneal cancer subjects must be newly diagnosed with epithelial ovarian cancer (stages II - IV), fallopian tube cancer with pelvic extension (stages II-IV), or primary peritoneal cancer (stages III-IV)
* Bladder, renal pelvis, or ureteral cancer subjects must be newly-diagnosed with muscle-invasive cancer (stages II - IV).
* Urethral cancer subjects must be newly diagnosed with cancer invading the corpus spongiosum, prostate, or periurethral muscle (stages II-IV)
* Subjects must be anticipated to receive chemotherapy without the concomitant treatment use of hormonal therapy or immunomodulators.

Exclusion Criteria:

* Subjects with other prior cancer diagnoses who have evidence of active disease
* Subjects who have received chemotherapy or radiation treatment within the past year (for any disease state)
* Subjects with melanoma or other non-squamous cell carcinoma of the head and neck
* Subjects with nasopharyngeal, sinonasal or lateral skull base tumors. Unintentional cranial irradiation can occur with treatment to these sites and could therefore not be completely eliminated from being associated with any cognitive deficits observed.
* Subjects with implanted non-MRI compatible metal objects, electrodes, pacemakers, intracardiac lines, or medication pumps
* Subjects with weight over 350 pounds (weight limit on MRI machine)
* Subjects with a history of claustrophobia
* Subjects with an inability to lie flat for 20 minutes (for fcMRI scan)
* Life expectancy of less than 6 months
* Any medical condition the Principal Investigator (PI) determines would not make the study safe or in the best interest of the potential subject to participate in.
* Subjects who receive hormonal therapy therapy or immunomodulators as part of their cancer therapy.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The final study population will include sixteen adults over the age of 40 years with newly-diagnosed locally-advanced breast, head and neck, ovarian, primary peritoneal, bladder , and urethral cancer although up to 25 patients will be approached for enrollment to account for losses to attrition.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2011-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in fcMRI | before and after chemotherapy
  Baseline and post-chemotherapy fcMRI maps will be compared for changes in degree of activation within the cognition-associated cortical networks. To compute statistical significance, correlation co-efficients from the fcMRI will be converted to a normal distribution using Fischer's r-to-z transformation.

SECONDARY OUTCOMES:
Correlation of change in fcMRI with change in neurocognitive test scores. | Baseline and at the completion of chemotherapy. Baseline visit must be no more than 2 weeks prior to start of chemotherapy. 2nd visit must occur within 2 weeks of last dose of chemotherapy.
  To assess the correlation between changes in cognition defined through standard neurocognitive tests and fcMRI among adult cancer patients after chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jay F Piccirillo, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States